CLINICAL TRIAL: NCT07110753
Title: The Effect of a Combined Lifestyle Intervention for Patients With Cancer on Quality of Life: the Randomized GLINK Study
Brief Title: The Effect of a Combined Lifestyle Intervention for Patients With Cancer on Quality of Life
Acronym: GLINK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Tilburg University (Other); VU University of Amsterdam (Other); Ede Christian University of Applied Sciences (Unknown)
Responsible Party: Principal Investigator, Kristel van Asselt, Epidemiologist and general practitioner, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NL-009215
Record Dates: First submitted 2025-06-25; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Cancer
Keywords: cancer; combined lifestyle intervention; quality of life; positive health
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Following a combined lifestyle intervention for 12 months
  Interventions: Behavioral: combined lifestyle intervention focusing on various lifestyle components, delivered by a lifestyle coach and oncology nurse
- Control group (Placebo Comparator): Receiving four online group sessions with a lifestyle coach and all educational materials after the intervention period of 6 months.
  Interventions: Behavioral: short online lifestyle intervention by lifestyle coach and educational materials after 6 months

INTERVENTIONS:
Behavioral: combined lifestyle intervention focusing on various lifestyle components, delivered by a lifestyle coach and oncology nurse — The combined lifestyle intervention focuses on various lifestyle components, including nutrition, physical activity, sleep, stress and sense of purpose, and is structured around the process of behaviour change. It is delivered by a lifestyle coach in collaboration with an oncology nurse.
  Arms: Intervention group
Behavioral: short online lifestyle intervention by lifestyle coach and educational materials after 6 months — The control group receives 4 online group sessions from a lifestyle coach and all educational materials after 6 months of intervention
  Arms: Control group

SUMMARY:
A growing number of people are living with the (long-term) consequences of cancer and its treatment, which can negatively affect their quality of life. This study aims to assess the effect of a combined lifestyle intervention for patients with cancer on quality of life.

DETAILED DESCRIPTION:
A growing number of people are living with the (long-term) consequences of cancer and its treatment, which can negatively affect their quality of life. The aim of this study is to assess the effect of a combined lifestyle intervention for patients with cancer, who suffer from the consequences of cancer and its treatment, on quality of life.

The GLINK study is a pragmatic randomized controlled trial with two study arms: an intervention (n=122)- and a control arm (n=122).

The investigators will recruit 244 cancer patients who have a reduced quality of life. Participants will be either within five years post-primary treatment OR have advanced cancer (stage IV) with a prolonged life expectancy. Patients in the intervention arm will be offered a combined lifestyle intervention guided by a lifestyle coach or oncology physiotherapist and oncology nurse. The intervention consists of an intensive intervention phase of 6 months and a maintenance phase of another 6 months. The control patients will receive four online group sessions with a lifestyle coach and all educational materials after the intervention period of 6 months.

The primary endpoint is quality of life. Secondary endpoints include Positive Health and lifestyle, various lifestyle changes and body measurements.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with an invasive or hematological cancer type and either within five years post-primary treatment with curative intent OR having advanced cancer (stage IV) with a prolonged life expectancy (chronic cancer patients) . Primary treatment in this context, includes among others surgery (> 3 months ago), radiotherapy, and/or chemotherapy or a stem cell transplant in case of hematological cancers.
* Report a reduced HRQoL, i.e., a low score on at least 2 of the functioning scales and/or the symptom scale fatigue of the EORTC-QLQ-30 based on the thresholds of clinical importance of Giesinger et al. (2020)
* Be 40 years of age or older. The investigators have chosen this cut-off because they believe that younger cancer patients (AYA's) face different challenges and should not be mixed with the average older patient. This approach ensures greater homogeneity within the study population.
* Be able to speak and understand Dutch

Exclusion Criteria:

* Following, or planned to follow a combined lifestyle intervention (i.e., one of the existing interventions for overweight) during the intervention period
* Patients in the terminal phase (life expectancy < 3 months)
* Mental or behavioural problems that hinder participating in group lifestyle coaching indicated by the health care professional who is referring to GLINK or by the study team
* Any circumstances that would impede ability to give informed consent or adherence to study requirements as determined by the study team or treating physician

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Health Related Quality of Life | Measured at 0, 6 and 12 months
  Summary score of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). This questionnaire consists of five functioning scales (physical, emotional, role, cognitive and social functioning), three symptom scales (fatigue, nausea & vomiting) and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The EORTC QLQ-C30 summary score ranges from 0 to 100, with higher scores indicating better health-related quality of life. This summary score is calculated as the mean of all scale scores (excluding global QoL and financial difficulties).

SECONDARY OUTCOMES:
Health-Related Quality of Life - separate functioning and symptom scales | Measured at 0, 6 and 12 months
  Separate functioning and symptom scales of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). This questionnaire consists of five functioning scales (physical, emotional, role, cognitive and social functioning), three symptom scales (fatigue, nausea & vomiting, and pain) and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). All scale and item scores range from 0 to 100. Higher scores on the summary score and function scales indicate a better quality of life. Higher scores on the symptom scales mean more symptoms.
Cancer-related fatigue | Measured at 0, 6 and 12 months
  Assessed with the Multidimensional Fatigue Inventory (MFI). The MFI is a 20-item questionnaire assessing five dimensions of fatigue: general, physical and mental fatigue, reduced activity, and reduced motivation. Each dimension has 4 items, and each item is scored on a 5-point Likert scale (1 to 5).The resulting scale scores for each dimension range from 4 to 20. Higher scores indicate higher levels of fatigue.
Sleep Hygiene | Measured at 0, 6 and 12 months
  Assessed with the Sleep Hygiene Index (SHI). The SHI is a questionnaire consisting of 12 items that assess sleep-related behaviors. The total score is the sum of all item responses, ranging from 0 to 52, with higher scores indicating worse sleep hygiene.
Positive Health | Measured at 0, 6 and 12 months
  Assessed with the 17-item Positive Health measurement tool, based on the Positive Health dialogue tool, which is widely used in the Netherlands. This tool measures six factors: physical fitness, mental functions, future perspectives, contentment, social relations, and health management. Items are scored on an 11-point scale ranging from 0 (totally disagree) to 10 (totally agree). For each factor, an average score can be calculated, with higher scores indicating better perceived Positive Health within that factor.
Height | Measured at 0 and 6 months
  Height (in centimeters) will be measured in light clothing without shoes using standardized procedures described in study SOPs.
Weight | Measured at 0 and 6 months
  Weight (in kilograms) measured in light clothing without shoes using standardized procedures described in study SOPS
Waist circumference | Measured at 0 and 6 months
  Waist circumference (in centimeters) will be measured in light clothing without shoes using standardized procedures described in study SOPs.
Body composition | Measured at 0 and 6 months
  To assess body composition (fat mass and fat free mass), a whole body bio impedance analysis will be performed at baseline and 6 months follow-up. Patients are measured in a lying position. Raw (i.e., reactance, resistance, and phase angle) or summary (fat (free) mass in kg) bioimpedance data are registered and for raw data estimates fat mass and fat-free mass are obtained using the Kyle equation.
Physical activity - questionnaire | Measured at 0, 6 and 12 months
  Assessed by the Short QUestionnaire to ASsess Health-enhancing physical activity (SQUASH). This questionnaire contains questions on commuting activities, leisure-time and sports activities, household activities, and activities at work. For each activity, participants report the number of days per week, the average duration per day (in minutes), and the perceived intensity (light, moderate, or vigorous). The outcomes are expressed in minutes of physical activity per week. Higher scores indicate a higher level of physical activity.
Physical activity - tracker | Measured at 0 and 6 months. The device will be worn for nine consecutive days, on the right mid-thigh, attached with adhesive tape.
  Assessed by the ActivPAL activity tracker (PAL technologies). The is small device, which has shown to reliable measure and distinguish between sitting time, standing time and stepping time.
Diet components | Measured at 0, 6 and 12 months
  Dietary related to cancer risk will be assessed: intake of fruit and vegetables, red and processed meat, and alcohol. These will be measured using items adapted from the Gezondheidsenquête CBS 2023 questionnaire, which is based on the Richtlijnen Goede Voeding 2015. Additionally, the use of nutritional supplements will be assessed.
Pack years of smoking | Measured at 0, 6 and 12 months
  Pack years (smoking duration * amount of cigartettes) will be assessed with a self-developed questionnaire.
Smoking status | Measured at 0, 6 and 12 months
  Smoking status (yes/no) will be assessed with a self-developed questionnaire.
Cost-effectiveness - EuroQol(EQ)-5D-5L | Measured at 0, 6 and 12 months
  The EuroQol 5-Dimensions 5-Levels (EQ-5D-5L) is used to measure health in five dimensions, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, using 5 levels of severity. The patients' EQ-5D-5L health states are converted into utility values using the Dutch tariff, after which they are used to calculate quality adjusted life years (QALYs).
Health care costs | Measured at 0, 6 and 12 months
  Assessed by a modified version of the iMTA Medical Cost Questionnaire (iMCQ)
Costs of Productivity loss | Measured at 0, 6 and 12 months
  Assesed by the Productivity Cost Questionnaire (iPCQ)
Costs of informal care | Measured at 0, 6 and 12 months
  Assessed by the iMTA Valuation of Informal Care Questionnaire (iVCQ)
Health literacy | Measured at 0, 6 and 12 months
  General health literacy will be measured with the Dutch Short Health Literacy Scale (HLS-EU-Q16). This questionnaire consists of three subscales: health care, disease prevention and health promotion. The B1-level translated Dutch version will be used. It consists of 16 items, each rated on a 4-point Likert scale ranging from 1 (very difficult) to 4 (very easy). Responses are dichotomized (1-2 = 0, 3-4 = 1) and summed into a total score ranging from 0 to 16, with higher scores indicating higher perceived health literacy.

CONTACTS AND LOCATIONS:
Overall Officials: Kristel van Asselt, PhD, MD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
The possibility of sharing individual participant data (IPD) will be determined at a later stage, taking into account applicable privacy regulations, ethical guidelines, and participant consent.

REFERENCES:
- See also: General website of the study where participants can find information and apply for the study.. — http://glinkstudie.nl